CLINICAL TRIAL: NCT06315998
Title: Accurate Identification of Structural Heart Disease Using Magnetocardiography as an Innovative and Non-invasive Tool
Brief Title: Diagnosis of Structural Heart Disease Using MCG
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: MCG-Structural
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-02

CONDITIONS: Structural Heart Abnormality
MeSH Terms: interventions — Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training and testing cohort
  Interventions: Device: Magnetocardiography
- External validation cohort
  Interventions: Device: Magnetocardiography

INTERVENTIONS:
Device: Magnetocardiography — Magnetocardiography

SUMMARY:
The purpose of this prospective cohort study is to determine the parameters of cardiac magnetic imaging to identify structural heart disease using use transthoracic echocardiography or cardiac magnetic resonance as reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Those with suspected structural heart disease who are scheduled to undergo echocardiography or cardiac magnetic resonance. Structural heart disease includes cardiomyopathy (hypertrophic cardiomyopathy, dilated cardiomyopathy, restrictive cardiomyopathy, etc.), congenital heart disease (including ventricular septal defect, atrial septal defect, patent ductus arteriosus, Tetralogy of Fallot) syndrome, tricuspid valve malformation, etc.), valvular heart disease (aortic valve stenosis, mitral valve stenosis, etc.), ventricular remodeling caused by myocardial ischemia or cardiac structural changes.
* Signed the consent form.

Exclusion Criteria:

* Those with atrial fibrillation, supraventricular tachycardia, atrioventricular block and other arrhythmias that have not returned to normal;
* Those who are thought to be incapable of completing the relevant examinations by an attending physicians (or physicians with higher qualifications) due to unstable clinical conditions, metal implants, etc., or those who are unable to perform the examinations;
* Those with obvious abnormal thyroid function, severe anemia or other blood diseases and other diseases that obviously affect the circulating blood supply;
* Those with malignant tumors;
* Pregnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected structural heart disease who are scheduled to undergo echocardiography or cardiac magnetic resonance
Sampling Method: Non-Probability Sample
Enrollment: 2914 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the MCG in identifying structural heart disease | from the date of enrollment until the date of discharge, up to 30 days
  Using echocardiography or cardiac magnetic resonance as reference standard to assess the sensitivity, specificity, accuracy, positive predictive value, negative predictive value, and ROC of the cardiac magnetic image algorithm model for identification and localization of structural heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- China, Shandong Qilu Hospital of Shandong University, Jinan, Shandong, China